CLINICAL TRIAL: NCT05830786
Title: Effectiveness of Virtual Reality in Orthopaedic Surgical Education: A Multistage Randomized Controlled Trial
Brief Title: Virtual Reality in Orthopaedic Surgical Education: A Randomized Controlled Trial
Acronym: VR-ORS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Robert Koucheki, Principal Investigator, Lead Researcher, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 44020
Record Dates: First submitted 2023-03-05; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Surgical Education; Virtual Reality; Orthopaedic Training
Keywords: Virtual Reality; Orthopaedic Training; Surgical Education; Head mounted display
MeSH Terms: interventions — Smart Glasses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors will be blinded to participant group allocation. Participants will also be blinded to group assignment up to the point of study initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive virtual reality (IVR) group (Experimental): The experimental group will experience various surgical training modules using immersive virtual reality.
  Interventions: Device: Immersive virtual reality (IVR)
- Traditional hands on orthopaedic workshop group (Active Comparator): Hands-on orthopaedic workshop sessions (including arthroscopy simulators, cadaveric models, and Sawbones®) in differing orthopaedic subspecialties (including sports, arthroplasty, and spine surgery).
  Interventions: Other: Traditional hands on orthopaedic workshop group

INTERVENTIONS:
Device: Immersive virtual reality (IVR) — Using Oculus Quest 2 (Reality Labs, Meta Platforms, United States) headsets the PrecisionOS platform version 3.0 (PrecisionOS Technology, Canada) virtual reality surgical modules will be utilized.
  Other Names: head mounted display; virtual reality
  Arms: Immersive virtual reality (IVR) group
Other: Traditional hands on orthopaedic workshop group — Hands-on orthopaedic workshop sessions (including arthroscopy simulators, cadaveric models, and Sawbones®) in differing orthopaedic subspecialties (including sports, arthroplasty, and spine surgery).
  Arms: Traditional hands on orthopaedic workshop group

SUMMARY:
Immersive virtual reality (IVR) surgical simulators are increasingly being used for learner education. The aim of this randomized controlled trial is to compare the efficacy of IVR to hands-on orthopaedic workshop sessions (such as arthroscopy simulators, cadaveric models, and Sawbones®) in various orthopaedic subspecialties (such as sports, arthroplasty, and spine surgery).

Overall, in this multi-stage comprehensive randomized controlled the aim is to assess:

1. If IVR simulation using head-mounted displays (HMD) is superior to the current standard of training for orthopaedic surgery residents and medical students.
2. Determine if it is feasible to incorporate immersive headset virtual reality simulation into residency training programs and medical school curriculums.
3. Assess the longitudinal application of IVR training on medical student and resident surgical education.

DETAILED DESCRIPTION:
Study Stages:

Stage 1 - Medical students and orthopaedic residents participating in the Canadian Orthopaedic Surgery Medical Education Course 2023 (COSMEC) will be selected and computer randomized (1:1) into two groups of experimental (IVR) and control (arthroscopy simulator box), based on level of training. Allocation concealment will be ensured using central randomization. Trainees in both groups will receive a common didactic training for knee arthroscopy. Subsequently, trainees in the experimental group will undergo a IVR surgical training module and trainees in the control group will undergo a similar module using arthroscopy simulator box. Following the training modules, participants will complete knowledge tests, technical skill assessments on knee arthroscopy simulators, and experiential surveys.

Stage 2 - Medical students and orthopaedic residents participating in the 2023 University of Toronto Orthopaedic Surgery bootcamp will be selected and computer randomized (1:1) into two groups of experimental (IVR) and control (sawbones), based on level of training. Allocation concealment will be ensured using central randomization. Trainees in both groups will receive a common didactic training for femoral intramedullary nail (IMN) placement. Subsequently, trainees in the experimental group will undergo a IVR surgical training module and trainees in the control group will undergo a similar module using Sawbones ®. Following the training modules, participants will complete knowledge tests, technical skill assessments on cadaveric models, and experiential surveys.

Stage 3 - The protocol explained in stage 1 and 2 may be repeated for various orthopaedic sub-speciality (including arthroplasty and spine surgery) for the participants in the booth camp.

Stage 4 - All trainees may then be followed longitudinally over the course 6 months. Trainees' performance may be evaluated for procedures in which training was provided, based on preceptor evaluations (for example by completing standardised evaluation forms) on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

* Being a University of Toronto medical student.
* Being a University of Toronto orthopaedic surgery resident.

Exclusion Criteria:

* Previous graduation from an orthopaedic surgery residency in Canada or abroad.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-16 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Objective Structured Assessment of Technical Skills (OSATS) | 2 weeks after the training sessions, over 30 minutes testing period
  The primary outcome of the study is to assess trainee procedural performance using simulators or cadaveric models between the experimental (IVR) and control groups, measured by Objective Structured Assessment of Technical Skill (OSATS) score.

SECONDARY OUTCOMES:
Global Ratings Scale (GRS) | 2 weeks after the training sessions, over 30 minutes testing period
  GRS will be used as a secondary outcome measure to evaluate the performance of the surgical trainees who will be participating in the study. The GRS scores will be recorded by expert evaluators who will observe the trainees performing the surgical procedure. The scores will be analyzed to assess the effect of the intervention on the overall performance of the trainees.
Hand and body motion analysis using sensors | 2 weeks after the training sessions, over 30 minutes testing period
  Motion analysis is used to evaluate the effectiveness of the training intervention and can help identify areas for improvement in surgical technique. By incorporating this objective measure, we can gain a more comprehensive understanding of the impact of the training interventions on surgical performance.
Experimental and confidence questionnaire | 2 weeks after the training sessions, over 30 minutes testing period
  Experimental and confidence questionnaire will be used to assess the participants' confidence level and perception of their own skills in performing the simulated laparoscopic task. This questionnaire will include questions regarding their comfort level with the equipment, confidence in their ability to complete the task accurately and efficiently, and their overall perception of their own skill level. The questionnaire will be administered after each simulation session and will be used to assess any changes in the participants' confidence and perception of their own abilities throughout the study. The results of this questionnaire will provide valuable insight into the participants' perceived skill level, and may be used to inform future training programs or interventions aimed at improving surgical skills.
Time to complete the procedure | 2 weeks after the training sessions, over 30 minutes testing period
  This secondary outcome will measure the total time required to complete the procedure, from the start of the procedure to the end. The time will be recorded in minutes using a stopwatch, and any breaks or interruptions during the procedure will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Wolfstadt, MD, Principal Investigator — University of Toronto; Peter Ferguson, MD, Principal Investigator — University of Toronto; Johnathan R Lex, MB ChB, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No
IPD is not going to be shared with other researchers. All participants' information will be de-identified. Participants are identified in research records only with a unique study identification number that is linked in a master code-breaking enrollment log. Aggregate data will be analyzed.